CLINICAL TRIAL: NCT04580043
Title: Experimental Manipulation of OFC Function and Behavioral Context: Towards an Integrative Translational Model of Compulsive Behaviors
Brief Title: Theta Burst Stimulation Plus Habit Override Training for Compulsive Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rebecca Price (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Rebecca Price, Associate Professor of Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY19090219 (Part 2); R01MH124707 (NIH)
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Compulsive Behavior; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Compulsive Behavior; Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- cTBS + Habit Override Training (Experimental): Transcranial Magnetic Stimulation delivered in a continuous Theta Burst Stimulation (cTBS) pattern, paired with Habit Override Training.
  Interventions: Behavioral: Habit Override Practice; Device: Transcranial Magnetic Stimulation
- Sham TBS + Habit Override Training (Active Comparator): Sham Transcranial Magnetic Stimulation, paired with Habit Override Training.
  Interventions: Behavioral: Habit Override Practice; Device: Sham Transcranial Magnetic Stimulation
- cTBS + Sham Training (Active Comparator): Transcranial Magnetic Stimulation delivered in a continuous Theta Burst Stimulation (cTBS) pattern, paired with Sham Training.
  Interventions: Device: Transcranial Magnetic Stimulation; Behavioral: Sham Training
- Sham TBS + Sham Training (Sham Comparator): Sham Transcranial Magnetic Stimulation, paired with Sham Training.
  Interventions: Behavioral: Sham Training; Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Behavioral: Habit Override Practice — Computerized "brain training" to provide practice in overriding avoidance habits.
  Arms: Sham TBS + Habit Override Training; cTBS + Habit Override Training
Device: Transcranial Magnetic Stimulation — Non-invasive method for temporary, focal stimulation of brain areas. Delivered in a continuous Theta Burst Stimulation (TBS) pattern.
  Other Names: cTBS
  Arms: cTBS + Habit Override Training; cTBS + Sham Training
Behavioral: Sham Training — Computer-based task practice in a non-active/inert task.
  Arms: Sham TBS + Sham Training; cTBS + Sham Training
Device: Sham Transcranial Magnetic Stimulation — Sham stimulation of non-brain areas. Delivered in a continuous Theta Burst Stimulation (TBS) pattern.
  Other Names: Sham cTBS
  Arms: Sham TBS + Habit Override Training; Sham TBS + Sham Training

SUMMARY:
This project seeks to identify causal neural mechanisms underlying unwanted, repetitive behaviors (compulsions). Using non-invasive brain stimulation coupled with practice in a computer task, we will modulate activity in a target brain region and measure effects on compulsive behaviors and related measures. This work could ultimately lead to the ability to treat compulsions more effectively by targeting the regions of the brain that can help or hinder attempts to overcome compulsions.

ELIGIBILITY:
Inclusion Criteria:

Participants will:

1. Be between the ages of 18 and 60 years
2. Endorse problematic compulsive behaviors, per self-report and clinician-administered measures.
3. Agree to video taping of structured clinical interview
4. Report that they will reside in the Pittsburgh area for at least 5 weeks

Exclusion Criteria:

1. Failure to meet standard MRI inclusion criteria: those who endorse claustrophobia, those who have cardiac pacemakers, neural pacemakers, surgical clips in the brain or blood vessels, surgically implanted metal plates, screws or pins, cochlear implants, implanted uterine devices, metal braces, or other metal objects in their body, especially in the eye. Dental fillings do not present a problem. Plastic or removable dental appliances do not require exclusion. History of significant injury or surgery to the brain or spinal cord that would impair interpretation of results. Pregnancy, determined by pregnancy tests on females.
2. Medical contraindications for Transcranial Magnetic Stimulation (TMS):

   1. Presence of a neurologic disorder or medication therapy known to alter seizure threshold (e.g., stroke, aneurysm, brain surgery, structural brain lesion, brain injury, frequent/severe headaches)
   2. Recurrent seizures or epilepsy in participant or family history of hereditary epilepsy
   3. Pregnancy
   4. Metallic implants in body or other devices that may be affected by magnetic field
   5. Significant heart disease or cerebrovascular disease
   6. Medications with strong seizure threshold lowering potential or which may interfere with the efficacy of TMS (e.g., clozapine, stimulants)
3. Acute suicidality or other psychiatric crises requiring treatment escalation
4. Changes made to treatment regimen within 4 weeks of baseline assessment
5. Reading level <6th grade as per participant self-report
6. Presence of bipolar, psychotic, autism spectrum, or substance use disorder (i.e. current problematic use of mood altering drugs such as cocaine, opiates, amphetamines, and barbiturates)
7. Presence of movement disorder or tics affecting manual responses
8. Inability to read text from 2 feet away (corrective lenses allowed)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Brain activation in target region | 10-60min post-intervention
  Mean Cerebral Blood Flow (CBF) in orbitofrontal cortex collected via functional Magnetic Resonance Imaging (fMRI)
Effort to resist compulsive behaviors in response to laboratory triggers | 60min post-intervention
  Custom-made laboratory assessment of ability to override compulsive behaviors in response to idiographic triggers: self-reported effort needed to resist (0-100 scale)
Duration of compulsive behaviors in response to laboratory triggers | 60min post-intervention
  Custom-made laboratory assessment of ability to override compulsive behaviors in response to idiographic triggers: duration of compulsive behavior performance (% of total time allotted)
Intensity of urges to perform compulsive behaviors in response to laboratory triggers | 60min post-intervention
  Custom-made laboratory assessment of ability to override compulsive behaviors in response to idiographic triggers: self-reported urge intensity (0-100 scale)

SECONDARY OUTCOMES:
Goal-directed cognition | 90min-1 week
  Neuropsychological test of flexible goal-directed cognition (two-step task): switch score (higher score=better performance)
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 1 week
  Clinician-administered measurement of obsessions and compulsions (range: 0-40; higher score=worse outcome)
WHO Disability Assessment Scale 2.0 | 1 week
  Self-report measure of general functioning and disability (0-100; higher score=worse outcome)
Obsessive Compulsive Inventory-Revised (OCI-R) | 1 week
  Self-report measure of obsessions and compulsions (0-72; higher score=worse outcome)
Effort to resist compulsive behaviors in response to laboratory triggers | 1 week
  Custom-made laboratory assessment of ability to override compulsive behaviors in response to idiographic triggers: self-reported effort needed to resist (0-100 scale)
Duration of compulsive behaviors in response to laboratory triggers | 1 week
  Custom-made laboratory assessment of ability to override compulsive behaviors in response to idiographic triggers: duration of compulsive behavior performance (% of total time allotted)
Intensity of urges to perform compulsive behaviors in response to laboratory triggers | 1 week
  Custom-made laboratory assessment of ability to override compulsive behaviors in response to idiographic triggers: self-reported urge intensity (0-100 scale)
Brain activation in target region | 1 week
  Mean Cerebral Blood Flow (CBF) in orbitofrontal cortex collected via functional Magnetic Resonance Imaging (fMRI)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca B Price, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT04580043/ICF_000.pdf